CLINICAL TRIAL: NCT00733642
Title: An Open Label, Single Dose Escalation Study Of PF-04360365 In Subjects With Mild To Moderate Alzheimer's Disease
Brief Title: Single Dose Escalation Study of PF-04360365 In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A9951008
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer's Disease
Keywords: antibody amyloid Alzheimer's Disease AD
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04360365 1 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 1 mg/kg
- PF-04360365 3 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 3 mg/kg
- PF-04360365 5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 5 mg/kg
- PF-04360365 10 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 10 mg/kg

INTERVENTIONS:
Biological: PF-04360365 1 mg/kg — PF-04360365 1 mg/kg infused as a single dose
  Arms: PF-04360365 1 mg/kg
Biological: PF-04360365 3 mg/kg — PF-04360365 3 mg/kg infused as a single dose
  Arms: PF-04360365 3 mg/kg
Biological: PF-04360365 5 mg/kg — PF-04360365 5 mg/kg infused as a single dose
  Arms: PF-04360365 5 mg/kg
Biological: PF-04360365 10 mg/kg — PF-04360365 10 mg/kg infused as a single dose
  Arms: PF-04360365 10 mg/kg

SUMMARY:
The purpose of this study is to determine whether single doses of PF-04360365 is safe and well tolerated in patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-child bearing potential) subjects ages ≥50 years of age.
* Diagnosis of probable AD (of mild to moderate severity), consistent with criteria from both: NINCDS-Alzheimer's Disease and Related Disorders Association (ADRDA) and DSM-IV-TR.
* MMSE score of 16-26 inclusive.
* Rosen-Modified Hachinski Ischemia Score ≤4.
* On a stable dose of background cholinesterase inhibitors or memantine for at least 60 days prior to dosing.

Exclusion Criteria:

* Diagnosis or history of other dementia or neurodegenerative disorders.
* Diagnosis or history of clinically significant cerebrovascular disease.
* Specific findings on magnetic resonance imaging (MRI); cortical infarct, micro hemorrhage, multiple white matter lacunes.
* History of allergic or anaphylactic reactions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To examine the safety and tolerability of a single dose of PF-04360365 in subjects with mild-to-moderate AD. | 6 months

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of PF-04360365 following administration of an IV infusion in subjects with mild-to-moderate AD. | 6 months
To evaluate the relationship of PF-04360365 plasma exposure and Aβ plasma exposure. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Eatontown, New Jersey
  - Pfizer Investigational Site, Oakhurst, New Jersey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951008&StudyName=Single%20Dose%20Escalation%20Study%20of%20PF-04360365%20In%20Subjects%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease